CLINICAL TRIAL: NCT01804920
Title: D-SERINE TREATMENT FOR TARDIVE DYSKINESIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herzog Hospital (Other)
Responsible Party: Principal Investigator, Heresco-Levi Uriel, Director - Psychiatry Department, Herzog Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1600
Record Dates: First submitted 2013-03-03; First posted 2013-03-05 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia and Schizoaffective Disorder; Tardive Dyskinesia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Tardive Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-serine adjuvant treatment (Experimental): Random assignment, parallel group, double blind, placebo controlled 8 weeks trial.
  First arm: D-serine adjuvant treatment, up to 4 g/day Second arm: Placebo adjuvant treatment
  Interventions: Dietary Supplement: D-serine
- Placebo adjuvant treatment (Placebo Comparator): Random assignment, parallel group, double blind, placebo controlled 8 weeks trial.
  First arm: D-serine adjuvant treatment, up to 4 g/day Second arm: Placebo adjuvant treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: D-serine
  Arms: D-serine adjuvant treatment
Dietary Supplement: Placebo
  Arms: Placebo adjuvant treatment

SUMMARY:
Presently no generally effective treatments for tardive dyskinesia (TD) are available. D-serine is a naturally occurring amino acid that acts in-vivo as positive allosteric modulator at the glycine site associated with the glutamatergic NMDA receptor. Previous studies have suggested that D-serine may improve motor symptoms, including dyskinesias, which are caused by treatment with presently used antipsychotics drugs.

The hypothesis under investigation in the present study is that D-serine adjuvant treatment may improve TD in schizophrenia patients diagnosed with this disorder.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-70;
2. diagnosis of schizophrenia/schizoaffective disorder according to DSM-IV criteria; diagnosis will be made on the basis of SCID interview and information from medical records, previous treating psychiatrists, and family informants;
3. history of ≥3 months antipsychotic drugs treatment and present stable dose antipsychotic treatment for at last 4 weeks;
4. fulfillment of Schooler-Kane TD research criteria on a first evaluation performed 2-12 weeks prior to study entrance and on a subsequent evaluation performed prior to allocation to experimental treatment.

Exclusion Criteria:

1. meeting criteria for other DSM-IV Axis I diagnoses;
2. presence of a neurological disorder or history of significant head injury;
3. substance abuse or alcoholism during entire lifetime;
4. are judged clinically to be at suicidal or homicidal risk;
5. female patients who are pregnant or lactating; female patients who are not pregnant or lactating, if sexually active, must be using medically accepted means of contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in AIMS total score | biweekly during a period of 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Heresco-Levy, MD, Principal Investigator — Herzog Hospital
Locations (1):
- Herzog Hospital, Jerusalem, Israel